CLINICAL TRIAL: NCT07302451
Title: REDI-CaP (Recovery of Erectile Dysfunction Induced in Prostate Cancer Patients). Innovative Management of Patients With Unfavorable Intermediate-Risk Prostate Cancer: a Special Focus on Quality of Life and Erectile Function Recovery
Brief Title: REDI-CaP(Recovery of Erectile Dysfunction Induced in Prostate Cancer Patients)
Acronym: REDI-CaP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Principal Investigator, Rossella Di Franco, Principal Investigator - Radiation Oncology, National Cancer Institute, Naples
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT IRCCS Fondazione Pascale; EUCT number: 2025-521170-33-00 (Other: Istituto Nazionale Tumori IRCCS Fondazione Pascale di Napoli)
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer (Adenocarcinoma)
Keywords: Erectile Function Recovery; Relugolix; Androgen Deprivation Therapy (ADT); Stereotactic Body Radiotherapy (SBRT); Cyberknife System; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — relugolix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unfavorable Intermediate-Risk Prostate Cancer (Experimental): This single arm study includes male patients over 18 years of age with histologically confirmed unfavorable intermediate-risk prostate cancer, defined as clinical stage T2b-T2c, PSA ≤ 20 ng/mL, Gleason score 7 (4+3), and ISUP grade 3. Participants must have a prostate volume < 80 cc, preserved erectile function (IIEF-5 > 8), ECOG performance status 0-1, and no evidence of capsular invasion or metastatic disease (based on multiparametric MRI, PSMA PET, CT with contrast, and bone scan).
  Interventions: Combination Product: Combined Androgen Deprivation Therapy with Relugolix and Image-Guided Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Combination Product: Combined Androgen Deprivation Therapy with Relugolix and Image-Guided Stereotactic Body Radiotherapy (SBRT) — Participants will receive oral androgen deprivation therapy (ADT) with Relugolix (120 mg daily for 12 months) and stereotactic body radiotherapy (SBRT) via CyberKnife®. ADT includes a neoadjuvant phase (months 1-3), concurrent SBRT phase (month 4), and adjuvant phase (months 5-12). About 7-10 days before SBRT, 3-4 intraprostatic fiducial markers will be implanted. SBRT consists of 5 fractions of 7.25 Gy (total 36.25 Gy) delivered over two weeks. Planning involves contrast-enhanced CT, with defined CTV and PTV, and sparing of organs at risk. Treatment uses real-time image guidance and motion tracking. The regimen aims to optimize tumor control while minimizing toxicity. Patients are monitored using RTOG criteria, quality of life questionnaires, PSA/testosterone levels, and financial toxicity assessments over an 18-month follow-up.

SUMMARY:
The goal of this study is to evaluate the recovery of erectile function at six months after hormonal therapy cessation in male patients affected by advanced prostate cancer and undergoing radiotherapy. The main questions are:

* How well and how quickly do patients recover their sexual function and overall quality of life after stopping hormone therapy and receiving radiotherapy?
* How do the details of the radiation treatment (like the dose and how it's delivered) relate to treatment success, side effects, and long-term outcomes such as cancer control, survival, and financial impact? Participants will receive hormonal therapy (Relugolix) following by radiotherapy. They will complete questionnaires on sexual function, quality of life, and financial impact before, during and after treatment, and attend follow-up visits for health assessments. The study will measure how many patients recover erectile function within six months of stopping hormonal therapy, how long recovery takes, how treatment doses relate to outcomes, and assess cancer control, side effects, quality of life, and survival.

DETAILED DESCRIPTION:
Assessment of the International Index of Erectile Function-5 (IIEF-5) score at six months after hormonal therapy cessation, indicating recovery in at least 70% of the study population. Evaluation of Erectile Function Recovery 6 Months After Hormonal Therapy Completion The success of the study will be determined if erectile function recovery is observed in at least 70% of the population 6 months after the completion of hormonal therapy. Definition of "Erectile Function Recovery" for Individual Patients: A subject will be considered to have recovered erectile function if, at 6 months after the completion of hormonal therapy (Relugolix), their IIEF5 (International Index of Erectile Function - 5) score meets one of the following conditions:

* Achieving an IIEF5 score ≥ 17: This score indicates mild erectile dysfunction or no erectile dysfunction (as per IIEF5 categories: 22-25 no erectile dysfunction, 17-21 mild dysfunction). AND/OR;
* Significant increase in IIEF5 score compared to baseline: An increase of at least 5 points compared to the baseline (pre-treatment) IIEF5 score, indicating a clinically significant improvement in erectile function.

Recovery will only be evaluated in patients who had erectile dysfunction present (IIEF5 < 22) at baseline. The study will be considered "successful" if the proportion of patients meeting the individual definition of "erectile function recovery" (as specified above) at 6 months after the completion of hormonal therapy is greater than or equal to 70% of the studied population.

The secondary endpoints of this study aim to provide a comprehensive understanding of both the functional and oncological outcomes following the cessation of hormonal therapy with Relugolix. One key endpoint is the time to sexual function recovery (SFRT), defined as the interval between hormonal therapy cessation and the point at which a patient achieves an IIEF-5 score of 8 or higher, maintained across two consecutive assessments. This threshold was selected to reflect a clinically meaningful level of erectile function recovery, particularly in patients with moderate to severe dysfunction at baseline, and aligns with established literature and the study's primary endpoint criteria. Recovery will be assessed by comparing post-treatment IIEF-5 scores with each patient's baseline value. Additionally, the study will investigate the correlation between erectile function recovery and radiation dose exposure to critical anatomical structures involved in sexual function, including the penile bulb, crura, internal pudendal arteries, periprostatic neurovascular bundles, and testes, aiming to identify dose-dependent effects on functional outcomes. Other secondary endpoints include biochemical progression-free survival (bPFS), measured according to the Phoenix criteria (nadir PSA + 2 ng/mL), as well as local control (time to local recurrence or last follow-up without recurrence) and distant progression-free survival (dPFS), defined as the time to detection of distant metastases. The study will also evaluate acute and late urinary and rectal toxicity, using the RTOG criteria and International Prostate Symptom Score (IPSS) to assess the genitourinary and gastrointestinal side effects of therapy. To gauge broader patient well-being, quality of life (QoL) will be monitored using validated tools including the EORTC QLQ-C30, EORTC PR25, and IIEF-5 questionnaires. Furthermore, the study incorporates a financial toxicity assessment using the PROFFIT questionnaire, which measures the economic burden of treatment from the patient's perspective. Lastly, overall survival (OS) will be tracked, defined as the time from treatment initiation to death from any cause or the date of last follow-up, thereby offering a complete view of treatment impact across survival, function, toxicity, and patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male sex. (This criterion is required for the patient population being studied and for the correct data structuring in CTIS.)
* Age > 18 years;
* Diagnosis of prostate cancer via transperineal core biopsy;
* Classified as unfavorable intermediate-risk (T2b-2c, PSA ≤ 20 ng/mL, and Gleason score 7(4+3); ISUP grade 3);
* Signed informed consent for REDI-CaP protocol;
* Signed consent for REDI-CaP data processing;
* Prostate volume < 80 cc;
* No evidence of prostate capsule invasion (documented by multiparametric MRI of the prostate);
* Performance status: 0-1;
* Negative total-body CT with contrast and bone scan for metastases;
* Negative PSMA PET for secondary lesions;
* IIEF-5 score: > 8;
* Patient compliance with completing periodic questionnaires and attending regular follow-ups as required by the study.

Exclusion Criteria:

* Have prostate cancer classified as low-risk, favorable intermediate-risk, or high-risk;
* Exhibit erectile dysfunction at baseline (IIEF-5 score: < 8);
* Show positive PSMA PET results for metastases or pelvic lymph nodes;
* Have capsular involvement documented by multiparametric prostate MRI;
* Have contraindications to radiotherapy and/or hormone therapy;
* Are unable to undergo MRI;
* Cannot adhere to periodic tests and follow-ups;
* Refuse or have contraindications to the implantation of intraprostatic fiducials.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Recovery of Erectile Function (IIEF-5) at 6 Months Post-ADT: ≥70% Threshold for Study Success | 6 months after completion of hormonal therapy (Relugolix)
  Assessment of erectile function recovery 6 months after cessation of hormonal therapy (Relugolix), using the International Index of Erectile Function-5 (IIEF-5). Recovery is defined as either (1) an IIEF-5 score ≥17 (indicating mild or no erectile dysfunction) and/or (2) an increase of ≥5 points from baseline. Only patients with baseline IIEF-5 <22 (i.e., some degree of erectile dysfunction) will be included in the analysis. The study will be considered successful if ≥70% of the eligible population meets the recovery criteria at the 6-month evaluation following ADT completion.

SECONDARY OUTCOMES:
Time to Sexual Function Recovery and Secondary Clinical Outcomes | From end of hormonal therapy to 36 months post-treatment
  Time from cessation of hormonal therapy to recovery of sexual function, defined as achieving and maintaining an IIEF-5 score ≥8 for at least two consecutive assessments. This threshold reflects clinically meaningful erectile function based on literature and the study's primary endpoint. Recovery will be evaluated relative to baseline. Correlations will be explored between recovery and radiation dose to critical structures (penile bulb, crura, internal pudendal artery, neurovascular bundles, testes). Additional outcomes include bPFS (Phoenix criteria), local control, dPFS, OS, urinary/rectal toxicity (RTOG, IPSS), QoL (EORTC QLQ-C30, PR25, IIEF-5), and financial toxicity (PROFFIT).

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Nazionale Tumori - IRCCS - Fondazione G. Pascale - Napoli, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No